CLINICAL TRIAL: NCT05677126
Title: A Randomized, Single-blind, Trial of Tralement Versus a Fixed-dose Trace Element Combination Product of Zinc, Copper, and Selenious Acid to Evaluate Manganese Safety in Pediatric Patients Requiring Long-term Parenteral Nutrition
Brief Title: Tralement vs. Fixed-dose Trace Element Combination Product in Patients >3 to 17 Years of Age Requiring Long-term PN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The Tralement Pediatric Safety Study has faced significant challenges in site recruitment and feasibility
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TE20002
Record Dates: First submitted 2022-12-13; First posted 2023-01-10 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-08

CONDITIONS: Manganese Safety in Pediatric Patients
MeSH Terms: interventions — Trace Elements; Zinc Sulfate; Copper Sulfate; manganese sulfate; Selenious Acid; Copper

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tralement (Active Comparator): This study will enroll new prescribed home parenteral nutrition users, i.e. a patient enrolled in the study within six weeks of initiating first-time use of long-term home parenteral nutrition requiring trace element additives. Note: a portion of patients who meet inclusion criteria may have received parenteral nutrition in an inpatient setting before discharge home.
  Interventions: Drug: Tralement
- a fixed-dose trace element combination product of zinc, copper, and selenious acid (Active Comparator): This study will enroll new prescribed home parenteral nutrition users, i.e. a patient enrolled in the study within six weeks of initiating first-time use of long-term home parenteral nutrition requiring trace element additives. Note: a portion of patients who meet inclusion criteria may have received parenteral nutrition in an inpatient setting before discharge home.
  Interventions: Drug: Fixed-dose trace element combination product of zinc, copper, and selenious acid

INTERVENTIONS:
Drug: Tralement — Tralement with Manganese
  Other Names: trace elements (zinc sulfate, cupric sulfate, manganese sulfate and selenious acid)
  Arms: Tralement
Drug: Fixed-dose trace element combination product of zinc, copper, and selenious acid — Tralement without Manganese
  Other Names: trace elements (zinc sulfate, cupric sulfate, manganese sulfate and selenious acid)
  Arms: a fixed-dose trace element combination product of zinc, copper, and selenious acid

SUMMARY:
Tralement versus a fixed-dose trace element combination product of zinc, copper, and selenious acid to evaluate product safety in pediatric patients >3 to 17 years of age requiring long-term parenteral nutrition.

DETAILED DESCRIPTION:
A Phase IV, multi-center, randomized single-blind trial to evaluate the safety profile of Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid in pediatric patients who are expected to require at least six-months of home parenteral nutrition.

This study will enroll new prescribed home parenteral nutrition users, i.e. a patient enrolled in the study within six weeks of initiating first-time use of parenteral nutrition requiring trace element additives. Note: a portion of patients who meet inclusion criteria may have received parenteral nutrition in an inpatient setting before discharge home.

Eligible participants who satisfy the inclusion requirements and no exclusion criteria will be consented to participate in this study and enter the screening study phase.

The screening evaluation will be conducted within 5 days of the dose administration of study drug. Study participants meeting entry criteria of normal brain MRI and laboratory manganese concentrations (whole blood/plasma/serum/RBC) will begin study drug on Day 1.

Participants will undergo 2 additional post-baseline brain MRI scans at Months 3 and 6 and have either 2 (3.5-<7 years of age) and 4 (7-16 years of age) separate neuropsychological tests at Day 1, Month 3, and Month 6. Additional clinical monitoring including safety and laboratory assessments will occur during the 6-month opt-in extension study.

All patients in each assigned trace element parenteral nutrition group will have parenteral nutrition formulations evaluated for manganese content at Day 1, Month 1, Month 3, and Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric (≥3 to 17 years of age) participants weighing >10 kg with assent to participation and his/her parent or legal guardian is willing and able to sign the informed consent approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC).
* Male and female participants who are new users to home parenteral nutrition as a source of trace elements when oral or enteral nutrition is not possible, insufficient, or, contraindicated.
* Anticipated duration of home parenteral nutrition use is 6 months or greater.
* A normal baseline brain MRI scan.
* A normal blood manganese concentration.
* Ability to undergo additional 2 brain MRI scans over the six-month study period (Sedation, if appropriate, to be determined by the Principal Investigator's study site, institutional review board recommendations, and parent/guardian assent).
* Definitive contraception for females of reproductive age.

Exclusion Criteria:

* Prior parenteral nutrition therapy.
* Hypersensitivity or allergy to zinc or copper.
* Baseline ferritin ≥300 ng/mL or below 100 ng/mL.
* Baseline Transferrin Saturation (TSAT) ≥45% or below 20%.
* Prior or current cholestatic liver disease defined as a clinical condition associated with decrease in bile flow due to impaired secretion by hepatocytes or to obstruction of bile flow through intra-or extrahepatic bile ducts.
* Liver function studies with transaminases greater than two-fold normal or total bilirubin >2 mg/dL.
* Brain MRI exclusion criteria: MRI-unsafe metal implants, claustrophobia.
* Known excess environmental exposure to manganese.
* Less than 1-year expected survival, as anticipated by their primary provider.
* Current participation in another clinical trial.
* Females in pregnant state.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of brain deposition of manganese in Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid. | Six months
  Change from baseline in basal ganglia index (BG-index) as determined by T1-weighted brain MRI images

SECONDARY OUTCOMES:
To assess the efficacy of Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid. | Six months
  Change from baseline in blood (plasma/serum/RBC) manganese levels
To assess the safety of Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid | Six months
  • Change from baseline in BG-index and pallidal index as determined by T1-weighted brain MRI images

OTHER OUTCOMES:
To assess efficacy of Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid for the subset of participants who are eligible to, and consent to, the extension study. | 12 months
  • Whole blood and plasma/serum/RBC manganese levels and other serum trace element levels
To assess the safety of Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid for the subset of participants who are eligible to, and consent to, the extension study. | 12 months
  • Change from baseline in BG-index and pallidal index as determined by T1-weighted brain MRI images

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, MD, Study Director — Medical Director